CLINICAL TRIAL: NCT03677557
Title: Safety, Tolerability, Patient Satisfaction and Cost of 16.5% Subcutaneous Immunoglobulin (Cutaquig®) Treatment in Patients Who Did Not Tolerate Other 20% Subcutaneous Immunoglobulin Product(s)
Brief Title: Safety, Tolerability, Patient Satisfaction and Cost of 16.5% Subcutaneous Immunoglobulin (Cutaquig®) Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018 0388-01H
Record Dates: First submitted 2018-07-06; First posted 2018-09-19 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Primary Immunodeficiency Disease; Secondary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cutaquig Intervention (Other): Participants with primary or secondary immunodeficiency disease who are currently on subcutaneous immunoglobulin treatment but have developed adverse events including allergic reaction and are willing to change the treatment product to 16.5% Cutaquig.
  Interventions: Drug: 16,5% Cutaquig

INTERVENTIONS:
Drug: 16,5% Cutaquig — Participants with primary or secondary immunodefiiciney disease and who do not tolerate other immunoglobulin treatments will be asked to use 16.5% Cutaquig

SUMMARY:
Patients with primary or secondary immunodeficiency disease who have developed adverse reactions to products available on the market such as Cuvitru® (Shire), Hizentra® (CSL Behring) or 10% Gammunex® (Grifols), may benefit from utilizing 16.5% Cutaquig® (Octapharma).

DETAILED DESCRIPTION:
This is a prospective interventional study before and after clinically driven change in treatment formulation.

Polyvalent immunoglobulin treatment is used in patients with primary or secondary antibody deficiency diseases to prevent and lower the risk of infection. There are multiple products available in the market. Most products are administered via intravenous route such as Privigen® (CSL Behring), Gammunex® (Grifols), and Panzyga® (Octapharma). Up until recently, there have been only two products that are licensed for subcutaneous administration - 20% Hizentra® (CSL Behring) and 10% Gammunex® (Grifols).

In our clinical experience, approximately 10% of patients treated with 20% Hizentra® developed adverse reactions. Some are mild and tolerable. Some are moderate to severe and required alteration of treatment plan: For example, changing the product from 20% Hizentra® to 10% Gammunex®. However, this results in a 100% increase in the injection volume due to the lesser concentration of the product, but a decrease in viscosity - both of which might alter overall tolerance. Likewise, any new treatment may bring new adverse events such as rash.

In 2018, there will be two additional subcutaneous immunoglobulin products available in Canada - 16.5% Cutaquig® (Octapharma) and 20% Cuvitru® (Shire).

Even though both new products are licensed and proven to be efficacious regarding preventing significant infection (1,2), the relative safety, tolerability, patient satisfaction, treatment-associated cost has not been studied in patients using the 16.5% Cutaquig®. The study product will be provided through the Canadian Blood Service (CBS) on a special request basis which is a standard procedure for any patients who are intolerable to inventory products.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients with primary or secondary immunodeficiency disease who are currently on subcutaneous immunoglobulin treatment but have developed adverse events and are willing to change the treatment product.

Exclusion Criteria:

* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events per participant per study visit of 16.5% Subcutaneous Immunoglobulin (Cutaquig®) Treatment | The outcome measure will be assessed through study completion, an average of 1 year
  The safety will be measured by the number of adverse events per participant per study visit
Retention of participants who are able to tolerate the study intervention at 12 months | Cumulative proportion of participants who are on Cutaquig at 12 months.
  Retention of participants who are able to tolerate the study intervention will be calculated as the number of participants enrolled between the 6 and 12 month visits
Quality of Life (Patient Satisfaction) | The outcome measure will be assessed through study completion, an average of 1 year
  This will be measured by quality of life questionnaire (SF-36) before and after change in treatment at 6 and 12 months
Patient satisfaction (Quality of life) | The outcome measure will be assessed through study completion, an average of 1 year
  This will be measured by quality of life questionnaire (Euroquol 5D-5L) before and after change in treatment at 6 and 12 months
Treatment associated cost | The outcome measure will be assessed through study completion, an average of 1 year
  This will measure the cost of nursing time and will be reported as dollars/patient/year

CONTACTS AND LOCATIONS:
Overall Officials: Juthaporn Cowan, MD, PhD, FRCPC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada